CLINICAL TRIAL: NCT05423769
Title: Safety and Effectiveness of Generic Fingolimod (Sphingomod®, Hikma) in Patients With Relapsing-Remitting Multiple Sclerosis in Egypt
Status: Completed | Type: Observational
Sponsor: Hikma Pharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: HIK-SPH-2021-01
Record Dates: First submitted 2022-06-14; First posted 2022-06-21 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-03

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: Fingolimod; Generic Fingolimod; Nervous System; Multiple Sclerosis; Relapsing-Remitting Multiple Sclerosis; Cohort Study; Observational Study; Effectiveness; Safety; Disease Modifying Treatments
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Neurologic Manifestations; Multiple Sclerosis | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Fingolimod — 0.5 mg hard gelatine capsules
  Other Names: Sphingomod®, Hikma

SUMMARY:
The purpose of this observational study is to evaluate the Safety and Effectiveness of Generic Fingolimod (Sphingomod®, Hikma) in Patients with Relapsing-Remitting Multiple Sclerosis in Egypt

DETAILED DESCRIPTION:
This is an observational, prospective, cohort study, where no visits or intervention(s) additional to the daily practice will be performed. In the study sites, patients undergoing routine clinical care for RRMS and initiating treatment with generic Fingolimod in accordance with the approved summary of product characteristics (SPC) will be followed up and assessed for a total of 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who initiate treatment with generic Fingolimod at baseline in accordance with the approved summary of product characteristics (SPC).
2. Males and females who are ≥ 18 years old.
3. Patients who had a diagnosis of RRMS per 2010 or 2017 revised McDonald criteria, who are:

   1. Newly diagnosed who had no prior Disease-Modifying Therapy (DMT), or
   2. Switched patients from Gilenya®, Novartis, or
   3. Switched patients from interferon beta (IFNβ).
4. Patients who agree to participate in the study and provide a written informed consent.

Exclusion Criteria:

1. Pregnant or lactating female patients and women of childbearing potential not using effective contraception.
2. Patients lacking immunity against varicella zoster virus (VZV).
3. Patients participating in other clinical studies.
4. Patients who meet any of the contraindications to the administration of the study drug according to the approved SPC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from different sites in Egypt
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with AEs and SAEs (including laboratory abnormalities). | up to 12 months from initiating generic Fingolimod.
Proportion of patients experiencing a relapse. | Time frame: up to 12 months period from initiating generic Fingolimod.
Time to First Relapse (TTFR) | up to 12 months from initiating generic Fingolimod.
Proportion of patients with disability progression as measured by the EDSS over time. | up to 12 months from initiating generic Fingolimod.

SECONDARY OUTCOMES:
Proportion of patients with AEs and SAEs (including laboratory abnormalities) leading to treatment discontinuation. | up to 12 months from initiating generic Fingolimod.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Neuropsychiatry department, Faculty of Medicine, Alexandria University Hospitals, Hadra University Hospital, Alexandria
  - Faculty of medicine Ain shams Research Institute-Clinical Research Center (MASRI-CRC), Cairo